CLINICAL TRIAL: NCT01976351
Title: Imaging Enhanced Endoscopy for the Screening of Barrett's Esophagus and Evaluation of Its Invasiveness in Patients With Gastroesophageal Reflux Disease
Brief Title: Imaging Enhanced Endoscopy for the Screening of Barrett's Esophagus
Status: Terminated | Type: Observational
Why Stopped: Insufficient research manpower
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200907036R
Record Dates: First submitted 2013-10-23; First posted 2013-11-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-10

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's esophagus; image-enhanced endoscopy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A standardized endoscopic biopsy protocol was performed at sites with ESEM which usually appeared as a reddish discoloration in an otherwise relatively whitish esophageal mucosa. Two pieces of specimen were taken; one for histological confirmation and another one (preserved as frozen tissue) for DNA analysis or immuno-histochemical staining. Biopsy from gastric cardia was also taken for histological confirmation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Barrett's esophagus: Patients were eligible for the study if they were scheduled for endoscopic examination at the National Taiwan University Hospital and its Yun-Lin branch, because of a BE, with or without a previous history of dysplasia. Exclusion criteria included patients who are younger than 20 years of age or patients with esophageal or cardiac varices or pregnant women.

SUMMARY:
Imaging enhanced endoscopy can improve the efficacy of screening of Barrett's esophagus and predict its invasiveness. There is potentially molecular change over the Barrett's esophagus in this Chinese population.

To evaluate the efficacy of imaging enhanced endoscopy for screening of Barrett's esophagus and evaluation of invasiveness

DETAILED DESCRIPTION:
Barrett ' s esophagus, defined as a pathological finding of metaplastic change of esophageal mucosa from squamous to columnar epithelium, is a tongue-like extension of salmon-colored mucosa from the gastroesophageal junction by endoscopy (1 2,3) . Endoscopic abnormalities suggestive of BE which has not been confirmed by histology, are defined as endoscopically suspected esophageal metaplasia (ESEM) (2). Barrett's esophagus is considered a precancerous lesion of esophageal adenocarcinoma (4 5) and it's mandatory for accurate diagnosis of BE. The pathogenesis of BE has also been closely associated with gastroesophageal reflux disease (6). In Western countries the reported prevalence of BE has varied from 0.9 to 4.5 % (3,7,8) in the general population and 6.3 to 13.6 % (9 - 12) in patients with GERD. For reliably rating differences of severity of endoscopically identified lesions among studies or quantify progression or regression of BE, International Working Group for the Classification of Oesophagitis (IWGCOA) proposed new classification of BE, the Prague C and M criteria (13) for defining the extent of BE based on the circumference (C) and maximum (M) of the lesion. This standard grading system could allow comparison of the severity of BE and aid in following the natural course of BE Image-enhanced endoscopy (IEE) compromises various means of enhancing contrast during endoscopy using dye, optical, and/or electronic methods IEE allows improved visualization of lesions and can be used to gain insight into the pathology of the lesion, Recent progress in optics and computerized processing of endoscopic images, such as narrow band image (NBI) and Fuji intelligent Chromoendoscopy (FICE), provide an optical and/or electronic enhancement of the mucosal structures. Most recently, the EPKi-processor (Pentax, Tokyo, Japan) developed i-Scan, a novel endoscopic post-processing light filter technology using delicate software algorithms with real-time image mapping technology, which can provide detailed analysis based on vessel (i-Scan V), pattern (i-Scan P), or surface architecture (i-Scan SE). Resolution of about 1.25 mega pixels per image could be provided by the computer-controlled digital processing. The SE-mode could be used for the identification of the morphological changes of esophageal mucosa. Accordingly, i-Scan e- and b-modes could be used to further evaluate the lesions, such as the regularity of vascular pattern and the presence of the abnormal vessels.

According to previous study (14), Ki67 and p53 immuno-histochemistry could reduce interobserver variation in assessment of Barrett's oesophagus. These IHC methods correlate with the severity of dysplasia very well and are useful supplementary prognostic markers In our study, we use the image enhanced endoscopy to observe the endoscopically suspected esophageal metaplasia and record it with Prague C and M criteria grading system. Immuno-histochemical staining was used as supplementary prognostic markers. Our aim is to evaluate the efficacy of imaging enhanced endoscopy for screening of Barrett's esophagus and evaluation of invasiveness.

ELIGIBILITY:
Inclusion Criteria:

* suspected or a history of Barrett's esophagus for endoscopic exam

Exclusion Criteria:

* younger than 20 years of age
* patients with esophageal or cardiac varices
* pregnant women.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were eligible for the study if they were scheduled for endoscopic examination at the National Taiwan University Hospital and its Yun-Lin branch, because of a BE, with or without a previous history of dysplasia. Exclusion criteria included patients who are younger than 20 years of age or patients with esophageal or cardiac varices or pregnant women.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The relationship between the mucosal morphology by imaging enhanced endoscopy and the presence of high-grade intraepithelial neoplasia from non-dysplastic specialized intestinal metaplasia. | Up to one month

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chia Lee, MD,Msc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan